CLINICAL TRIAL: NCT06540911
Title: Personalized Physical Back Training Program to Improve Physical Functioning in People with Non-specific Low Back Pain: a Feasibility Study
Acronym: LIFDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Luzern (Other)
Collaborators: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-01284; 63674 (Other Grant/Funding Number: Stiftung Universität Luzern)
Record Dates: First submitted 2024-07-19; First posted 2024-08-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Exercise Therapy; Exercise; Low Back Pain
Keywords: Exercise; Low Back Pain; Physical Functioning
MeSH Terms: conditions — Motor Activity; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized physical back training program (Experimental): 4-week personalized physical back training program
  Interventions: Other: Personalized physical back training program
- Non-personalized physical back training program (Active Comparator): 4-week non-personalized physical back training program
  Interventions: Other: Non-personalized physical back training program

INTERVENTIONS:
Other: Personalized physical back training program — The study intervention is a 4-week personalized physical back training program. The study intervention consists of six exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are selected through a clinical reasoning process, i.e., they are tailored and problem-oriented, based on the results of a clinical assessment.
  Arms: Personalized physical back training program
Other: Non-personalized physical back training program — The control intervention is a 4-week non-personalized physical back training program. The control intervention consists of six exercises selected from a predefined set by a physical therapist or medical doctor. These exercises are not selected through a clinical reasoning process, i.e., they are neither tailored nor problem-oriented nor based on the results of a clinical assessment.
  Arms: Non-personalized physical back training program

SUMMARY:
The aim of our clinical trial (2024-01285) is to determine how an individualized physical back training program affects physical functioning and back pain. The results will help identify the most effective treatments for low back pain. This feasibility study (2024-01284) aims to conduct a test run of the clinical trial. The main questions are:

* Do all procedures run smoothly?
* Does the back training program improve physical functioning?
* Does the back training program reduce back pain?

Participants will:

* Follow a back training program for 4 weeks.
* Attend group exercise sessions (30 minutes per week)
* Perform exercises at home (3x10 minutes per week).
* Fill out a daily questionnaire on pain and exercise adherence.

ELIGIBILITY:
Inclusion Criteria: Individuals who

* have access to the University Sports of the Lucerne Universities (i.e., students, employees, alumni, subscribers),
* report NSLBP for at least 6 weeks (e.g., no upper limit of pain duration),
* report activity limiting NSLBP (i.e., at least one activity with a PSFS Score of ≤ 5/10 on a scale from 0 = unable to perform due to NSLBP to 10 = able to perform at the same level as before NSLBP),
* identify NSLBP as their primary musculoskeletal complaint,
* are between 18 and 65 years of age,
* understand the German language,
* are willing to participate in the study (i.e., adhere to a 4-week intervention),
* and provide written informed consent.

Exclusion Criteria: Individuals who …

* have been diagnosed with specific LBP (e.g., fractures, carcinoma, anomalies, nerve root affection with neurological signs such as sensitivity or reflex loss, muscle weakness, or radicular pain below the knee),
* report red flags associated with any serious pathology or specific LBP (e.g., major trauma of the back, unintended weight loss, saddle anaesthesia, changes in bowel or bladder function associated with LBP, progressive lower extremity neurologic deficits, fever),
* are less than 12 months post-surgery following any surgery on the lower back,
* are on a waiting list for any surgery on the lower back,
* are pregnant or have given birth within the last 12 months,
* are planning to become pregnant in the next 12 months,
* have diagnosed peripheral and/or central neurological disease,
* have diagnosed psychological and/or psychiatric condition,
* have diagnosed chronic toxic substances abuse (i.e., drugs, alcohol),
* take specific medication (i.e., neuroleptics, sedatives, anti-epileptics, antidepressants),
* are not allowed to exercise during the intervention period (e.g., on medical advice, due to a health-related condition),
* or are expecting to be absent more than 2 weeks during the training intervention period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Logistical and operational feasibility: Response time | Baseline
  Response time (in days).
Logistical and operational feasibility: Recruitment capability | Baseline
  Ratio of invited individuals to included participants.
Logistical and operational feasibility: Sample characteristics | Baseline to 4 weeks
  Analyze sample characteristics (e.g., gender, age) using descriptive statistics.
Logistical and operational feasibility: Data collection procedures (Access) | Baseline to 4 weeks
  Qualitatively evaluate the access of study personnel to necessary documents and the database through interviews.
Logistical and operational feasibility: Data collection procedures (Questionnaire) | Baseline to 4 weeks
  Qualitatively evaluate the usability of the questionnaire through interviews.
Logistical and operational feasibility: Data collection procedures (Clinical Assessment) | Baseline to 4 weeks
  Qualitatively evaluate the usability of the clinical assessment through interviews.
Logistical and operational feasibility: Acceptability and suitability of the intervention and study procedures | Baseline to 4 weeks
  Qualitatively assess the acceptability and suitability of the intervention and study procedures through interviews.
Logistical and operational feasibility: Resource management | Baseline to 4 weeks
  Qualitatively evaluate the time and personnel required for conducting the study through interviews.

SECONDARY OUTCOMES:
Self-rated physical functioning (PSFS) | Baseline to 4 weeks
  Change in Patient-specific Functional Scale (PSFS), most bothersome activity. Range from 0 (unable to perform due to NSLBP) to 10 (able to perform at the same level as before NSLBP).
Self-rated physical functioning (RMDQ) | Baseline to 4 weeks
  Change in Roland Morris Disability Questionnaire (RMDQ). Range from 0 (no disability) to 24 (maximum disability).
Health-related quality of life (EQ-VAS) | Baseline to 4 weeks
  Change in EQ Visual Analogue Scale (EQ-VAS). Range from 0 (lowest health-related quality of life) to 100 (highest health-related quality of life).
Health-related quality of life (EQ-5D-5L) | Baseline to 4 weeks
  Change in 5-Level EuroQoL5D version (EQ-5D-5L). Range from 0 (lowest health-related quality of life) to 1 (highest health-related quality of life).
Pain intensity (NRS) | Baseline to 4 weeks
  Change in pain intensity (11-point Numeric Rating Scale, NRS). Range from 0 (no pain) to 10 (pain as bad as you can imagine). Recall period: 7 days.
Intervention-related (serious) adverse events | During the 4 week intervention period
  Number of serious adverse events (SAE) and adverse events (AE) that are deemed possibly, probably, or definitely related to the intervention (according to ClinO, Art. 63, Switzerland).

OTHER OUTCOMES:
Pain frequency | Baseline to 4 weeks
  Change in number of episodes with NSLBP. Numerically, with 0 = minimum. Recall period: 7 days.
Pain duration | Baseline to 4 weeks
  Change in pain duration (e.g., average duration of an episode of NSLBP within the last 7 days). In minutes, hours, or days, with 0 = minimum. Recall period: 7 days.
Pain interference (PEG) | Baseline to 4 weeks
  Change in Pain, Enjoyment, and General Activity (PEG) 3-Item Scale. Range from 0 (no pain; does not interfere) to 10 (pain as bad as you can imagine; completely interferes). Recall period: 7 days.
Pain extent | Baseline to 4 weeks
  Change in pain extent. Percentages of the body with NSLBP, with 0%=minimum
Performance-based physical functioning (pressure pain threshold) | Baseline to 4 weeks
  Change in pressure pain threshold. kPA, with 0=minimum
Performance-based physical functioning (range of motion) | Baseline to 4 weeks
  Change in range of motion. Degrees, with 0=minimum
Performance-based physical functioning (strength) | Baseline to 4 weeks
  Change in strength. Nm, with 0=minimum
Performance-based physical functioning (neurodynamics) | Baseline to 4 weeks
  Change in neurodynamics. Positive, negative.
Performance-based physical functioning (movement control) | Baseline to 4 weeks
  Change in movement control. Positive, negative.
NSLBP-related work productivity loss | Baseline to 4 weeks
  Change in Work Productivity and Activity Impairment Questionnaire (WPAI). Percentages, with 0%=no work productivity loss.
Participant satisfaction | Baseline to 4 weeks
  Change in participant satisfaction (e.g., 1) I am satisfied with the training program I received. 2) I am satisfied with the result of the training program). 5-point Likert scale (strongly agree, agree, uncertain, disagree, strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, Prof., Principal Investigator — University of Lucerne, Faculty of Health Sciences and Medicine, Universitäres Forschungszentrum Gesundheit und Gesellschaft, Frohburgstrasse 3, 6002 Luzern
Locations (1):
- University of Lucerne, Faculty of Health Sciences and Medicine, Universitäres Forschungszentrum Gesundheit und Gesellschaft, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to make encrypted individual participant data (IPD) available through a repository and/or via publications, such as supplementary materials
Supporting Information: Study Protocol
Time Frame: Data will be available from the completion of the study for at least 10 years.
Access Criteria: Access to the data will be granted according to the repository and/or publisher's criteria.